CLINICAL TRIAL: NCT02935556
Title: Characterization and Epigenetics of Post-Partum Preeclampsia
Status: Terminated | Type: Observational
Why Stopped: Low Accrual
Sponsor: Duke University (Other)
Collaborators: New York University (Other); Society for Obstetric Anesthesia and Perinatology (Other)
Responsible Party: Sponsor
Other Study IDs: PRO00104636
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Post Partum Pre-eclampsia
Keywords: Post Partum Pre-eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be isolated from the whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- post partum pre-eclampsia: women with normal deliveries followed by post partum pre-eclampsia within 1 month of delivery.
  Interventions: Other: no intervention
- controls: women with normal deliveries and normal post part courses who match the post partum pre-eclampsia women in age, BMI, smoking status, gestational age and race/ethnicity.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — database and epigenetic study

SUMMARY:
This study will recruit women with post partum pre-eclampsia and match them to controls without postpartum pre-eclampsia to identify an epigenetic signature that is specific to women with post partum pre-eclampsia to help characterize the underlying pathophysiology of post partum pre-eclampsia.

DETAILED DESCRIPTION:
Preeclampsia (PEC) is a heterogeneous disease that complicates 5-8% of pregnancies. Approximately 10% of PEC patients will present with post-partum PEC without having developed the syndrome during the pregnancy (PP-PEC). Management of post-partum preeclampsia (PP-PEC) is challenging because many women do not seek care until neurologic symptoms result from severe-range elevated blood pressure. The pathogenesis and clinical characteristics of PP-PEC are understudied and poorly understood. Identifying clinical risk factors and biomarkers of PP-PEC would help to identify women at risk.

ELIGIBILITY:
Inclusion Criteria:

* Post partum pre-eclampsia

Matching based on:

* maternal age (years +/-3)
* BMI (+/-5 points)
* Ethnicity
* Mode of delivery
* Gestational age at delivery (+/7 days)
* Smoking status

Exclusion Criteria:

* Intrapartum pre-eclampsia

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who present to the hospital with postpartum pre-eclampsia are matched with women who never have PP-PEC (post-partum preeclampsia).
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
methylation signature on circulating monocytes | 1 week post delivery

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Louise Meng, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No